CLINICAL TRIAL: NCT06715228
Title: Efficacy of Shitali Respiratory Rehabilitation Program in Obstructive Sleep Apnea
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, Department of Physical Therapy for Cardiovascular/Respiratory Disorder and Geriatrics, Faculty of Physical Therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00014233-15
Record Dates: First submitted 2024-11-28; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group I (Experimental): in this group, patients (n=20) with obstructive sleep apnea will participate and will administer six cycles of 5-min shitali respiratory pranayama exercise rehabilitation training (the rehabilitation will be repeated or applied at morning, afternoon, and also at evening) for 12 week as a daily performance,
  Interventions: Behavioral: shitali pranayama respiratory rehabilitation training
- Group II (No Intervention): in this group, patients (n=20) with obstructive sleep apnea will participate and will act as control group. In this group, no intervention will be applied

INTERVENTIONS:
Behavioral: shitali pranayama respiratory rehabilitation training — in this group, patients (n=20) with obstructive sleep apnea will participate and will administer six cycles of 5-min shitali respiratory pranayama exercise rehabilitation training (the rehabilitation will be repeated or applied at morning, afternoon, and also at evening) for 12 week as a daily performance
  Arms: group I

SUMMARY:
obstructive sleep apnea has a negative impact on blood pressure of patients, sleeping quality, and respiration

DETAILED DESCRIPTION:
in this study, patients (n=40) with obstructive sleep apnea will participate in this study to be divided in to group I and group II with an equal number of patients (n = 20 for the group). Group I will administer six cycles of 5-min shitali respiratory pranayama exercise rehabilitation training (the rehabilitation will be repeated or applied at morning, afternoon, and also at evening) for 12 week as a daily performance, the other group, Group II, will act as control group.

ELIGIBILITY:
Inclusion Criteria:

* non-obese patients
* obstructive sleep apnea (mild and moderate form)

Exclusion Criteria:

* cardiac patients metabolic diseases kidney diseases

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — based on self-representation of gender identity.
Enrollment: 40 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
apnea hypopnea index | it will be assessed after 12 weeks
  it will be measured through a sleep study

SECONDARY OUTCOMES:
systolic blood pressure | it will be assessed after 12 weeks
  it will be assessed via a sphygmomnamoeter
diastolic blood pressure | it will be assessed after 12 weeks
  it will be assessed via a sphygmomnamoeter
Pittsburg sleep quality index | it will be assessed after 12 weeks
  it will assess sleep quality
respiratory rate | it will be assessed after 12 weeks
  it will assess respiratory cycle per minute
Epworth sleepiness scale | it will be assessed after 12 weeks
  it ill assess daytime sleepiness
visual analogue scale of by-partner reported sleep difficulty | it will be measured after 12 weeks
  it will assess by-partner reported sleep difficulty due to snoring of patient

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ismail, lecturer, Principal Investigator — Cairo University
Locations (1):
- faculty of physical therapy Cairo university, Dokki, Giza Governorate, Egypt